CLINICAL TRIAL: NCT04150211
Title: Effects of Dietary Supplementation With Exten(d) Blend on Training Ability in Recreational Runners: A Pilot Randomized, Triple-blind, Placebo Controlled Trial
Brief Title: Effects of Exten(d) Supplementation on Training Ability in Recreational Runners
Acronym: Exten(d)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Natural Origins (Industry)
Collaborators: Universidad Politecnica de Madrid (Other)
Responsible Party: Principal Investigator, Marcela González-Gross, Proffessor Doctor, Universidad Politecnica de Madrid
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Nat.Origins-Exten(d)-2019
Record Dates: First submitted 2019-10-16; First posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Joint Pain; Knee Inflammation; Biomechanical; Lesion
Keywords: Harpagophytum; Zingiber officinae; Bixa orellana; Joint pain; Inflammation; Biomechanics
MeSH Terms: conditions — Arthralgia; Inflammation

STUDY DESIGN:
Intervention Model Description: Single dose, Randomized, triple Blinded, Placebo-controlled Study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Each pill bottle was assigned a five characters numeric code and a letter (A or B). Then, the codes were randomly distributed to the participants. Once the study finished, an external person to the study revealed the placebo and controlled group for each letter.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exten(d) (Active Comparator): Subjects have to take Exten(d) capsules (3 times a day, total 2 g/day) during breakfast, lunch and diner, during 4 weeks.
  Interventions: Dietary Supplement: Polyherbal Exten(d) vs Placebo
- Placebo (Placebo Comparator): Subjects have to take Placebo capsules (3 times a day, total 2 g/day) during breakfast, lunch and diner, during 4 weeks.
  Interventions: Dietary Supplement: Polyherbal Exten(d) vs Placebo

INTERVENTIONS:
Dietary Supplement: Polyherbal Exten(d) vs Placebo — Supplementation during 4 weeks

SUMMARY:
The study will assess running biomechanics and joint inflammation of physically active males between 40 and 60 years of age, mainly runners, suffering from knee joint inflammation and pain after training. Participants were split into two groups, intervention and placebo, to evaluate the safety and efficacy of Exten(d) supplementation during 4 weeks.

DETAILED DESCRIPTION:
Triple-blind, randomized, placebo-controlled, parallel group, pilot safety, and efficacy study.

30 healthy physically active males (40 to 60 years old) suffering from knee joint inflammation and pain after training were randomly assigned to the Exten(d) or Placebo group. During the first visit and after 4 weeks supplementation (either 2 g daily of Exten(d) capsules or placebo capsules) the participants were subjected to a three-stage exercise session: (i) running biomechanical assessment, (ii) exercise physiology maximal effort test and (iii) running biomechanical assessment after the incremental exercise to exhaustion. The volunteers have been assessed to determine: (1) inflammation by I-R thermography and pain perception, (2) running technics though biomechanic analysis and (3) performance.

ELIGIBILITY:
Inclusion Criteria:

* Male recreational runners who run for at least 150 minutes per week divided into two or more sessions.
* The participants were expected to describe some degree of knee inflammation and/or discomfort after training in order to be accepted. Knee discomfort was considered significant whenever a subject referred to a punctuation of ≥ 2 in a Visual Analogue Scale (VAS).
* Agree not to initiate any new exercise or diet programs during the entire study period
* Agree not to change their current diet or exercise program during the entire study period
* Agree not to stretch, utilize ice massage, take anti-inflammatory medications (eg, aspirin, ibuprofen), or use any other treatment during the trial.

Exclusion Criteria:

* Use of anti-inflammatory medications or pain medications 1 week before the screening visit and during the study
* Daily use of dietary supplements and herbal supplements beginning at the screening visit and during the study
* Antibiotic use in the past 3 months
* Chronic disease

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Effects of Exten(d) herbal blend on knee and popliteus inflammation | Changes from baseline at week 4
  Knee and popliteus inflammation assessment by IR Thermography after the warm-up, after the first Biomechanical test, after the incremental test to exhaustion and after the second biomechanical test.
Effects of Exten(d) on biomechanicals running technique | Changes from baseline running technique at week 4
  Biomechanics techniques assessment by VICON technology before and after the incremental test to exhaustion

SECONDARY OUTCOMES:
Enzymes safety variables | Changes from baseline at week 4
  Blood based biomarkers assay for liver injury enzymes (Alanine transaminase GPT, Aspartate transaminase GOT, Gamma glutamyl-transpeptidase GGT) and muscle injury CPK (IU/L)
Impedancemetric variables | Changes from baseline at week 4
  Body composition assessment (DXA): fat mass, lean mass, total water (%), muscle mass (kg)
VO2max | Changes from baseline at week 4
  VO2max assessment during an incremental test to exhaustion on a computerized treadmill. Expired gases measurment by a Jaeger Oxycon Pro gas analyser during the incremental test
knee pain perception | Changes from baseline at week 4
  Visual Analogue Scale pain perception
Biochemical variables | Changes from baseline at week 4
  Changes in metabolic biomarkers: total Bilirubin, Urea, Albumin, Creatinin, Cholesterol, HDL, LDL, TG
Hematological variables | Changes from baseline at week 4
  Changes in the hematological profile

CONTACTS AND LOCATIONS:
Overall Officials: Marcela Gonzalez-Gross, phD, Principal Investigator — INEF- Universidad Politecnica de Madrid
Locations (1):
- Universidad Politecnica de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalez-Gross M, Quesada-Gonzalez C, Rueda J, Sillero-Quintana M, Issaly N, Diaz AE, Gesteiro E, Escobar-Toledo D, Torres-Peralta R, Roller M, Guadalupe-Grau A. Analysis of Effectiveness of a Supplement Combining Harpagophytum procumbens, Zingiber officinale and Bixa orellana in Healthy Recreational Runners with Self-Reported Knee Pain: A Pilot, Randomized, Triple-Blind, Placebo-Controlled Trial. Int J Environ Res Public Health. 2021 May 22;18(11):5538. doi: 10.3390/ijerph18115538. PMID 34067240